CLINICAL TRIAL: NCT00941083
Title: Pilot, Open-label, Randomized, Single-center Study to Asses a Simplification Strategy From Protease Inhibitors to Raltegravir: Once Daily Isentress (ODIS)
Brief Title: Simplification From Protease Inhibitors to Raltegravir
Acronym: ODIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Carlos III, Madrid (Other)
Responsible Party: Hospital Carlos III, Vicente Soriano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC0509
Record Dates: First submitted 2009-07-14; First posted 2009-07-17 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: HIV Infections
Keywords: Simplification from protease inhibitors to raltegravir; Treatment Experienced; HIV-1 Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RAL QD 800 mg/24 hs (Experimental)
  Interventions: Drug: Raltegravir (Use RAL as a simplification strategy)
- RAL BID 400 mg/12 hs (Active Comparator)
  Interventions: Drug: Raltegravir (Use RAL as a simplification strategy)
- RAL BID to QD (Experimental)
  Interventions: Drug: Raltegravir (Use RAL as a simplification strategy)

INTERVENTIONS:
Drug: Raltegravir (Use RAL as a simplification strategy) — RAL QD: RAL 800 mg/24 hs
  Arms: RAL QD 800 mg/24 hs
Drug: Raltegravir (Use RAL as a simplification strategy) — RAL BID 400 mg/12 hs
  Arms: RAL BID 400 mg/12 hs
Drug: Raltegravir (Use RAL as a simplification strategy) — RAL BID to QD
  Arms: RAL BID to QD

SUMMARY:
A switch from protease inhibitors (PIs) to raltegravir (RAL) will be effective virologically and immunologically. Moreover, it will be associated with significant improvements in the lipid profile in HIV patients with undetectable viremia on PIs. In this setting, RAL once a day (QD) will perform as well as RAL twice a day (BID).

ELIGIBILITY:
Inclusion Criteria:

* HIV1 sero-positive using standard diagnostic criteria
* Plasma viral HIV-RNA below 50 copies/ml within 180 days prior to randomization
* On therapy with protease inhibitors both ritonavir-boosted or un-boosted for at least 6 months prior to study entry

Exclusion Criteria:

* Pregnancy or breast feeding
* Prior use of Integrase inhibitors
* Alcohol or substance abuse if according to the investigator opinion would interfere with compliance
* UIse of investigational medications within 30 days before study entry or during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with plasma HIV-RNA < 50 copies/ml at week 24 in each arm (RAL QD, RAL BID, RAL BID to QD) | 24 weeks

SECONDARY OUTCOMES:
CD4 gains, lipid profile, adverse events, | 24 weeks
Drug resistance mutations | 24 weeks
Raltegravir through plasma levels and correlation with virological failure | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Soriano, Dr, Principal Investigator — Hospital Carlos III
Locations (1):
- Hospital Carlos III, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Vispo E, Barreiro P, Maida I, Mena A, Blanco F, Rodriguez-Novoa S, Morello J, Jimenez-Nacher I, Gonzalez-Lahoz J, Soriano V. Simplification from protease inhibitors to once- or twice-daily raltegravir: the ODIS trial. HIV Clin Trials. 2010 Jul-Aug;11(4):197-204. doi: 10.1310/hct1104-197. PMID 20974575